CLINICAL TRIAL: NCT00154037
Title: Characterization of Vascular Effects of Candesartan and Pioglitazone.
Brief Title: Investigation of Vascular Relaxing Effects of Candesartan and Pioglitazone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IKPD 02-05
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Healthy Subjects
Keywords: vascular reactivity; venodilation; pulse wave velocity
MeSH Terms: interventions — Pioglitazone; Pharmaceutical Preparations; candesartan

INTERVENTIONS:
Drug: Pioglitazone (drug) and/or candesartan (drug)

SUMMARY:
The study is designed to test the hypothesis in healthy subjects that candesartan and pioglitazone provide additional vascular relaxing or modulating effects in addition to their blood-pressure and blood glucose level reducing ability, respectively.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of oral candesartan and/ or rosiglitazone therapy on the vascular responsiveness of different vasoactive compounds (angiotensin II, insulin, histamine and glyceroltrinitrate) in healthy subjects. Pioglitazone will be given orally (4 weeks 30mg/d, titrated to 45 mg/d for another 4 weeks). Candesartan will be given orally (4 weeks 8mg/d, titrated to 16 mg/d for another 4 weeks) as treatment. Every subject will receive intravenous stimulation with phenylephrine, angiotensin II, histamine, insulin and glyceroltrinitrate before and after an 8 weeks treatment interval with study medication or placebo. In addition, pulse wave velocity will me measured non-invasively before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male
* healthy
* 18 - 40 years old
* non-smoker
* no additional medication

Exclusion Criteria:

* any relevant disease
* smokers
* elevated liver enzymes
* body weight different from Broca Norm > 20%
* allergies

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-10; Study Completion 2006-09

PRIMARY OUTCOMES:
Vascular reactivity

SECONDARY OUTCOMES:
Pulse wave velocity
Changes in Angiotensin metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Kirch, MD, Study Chair — Institute of Clinical Pharmacology
Locations (1):
- Institute of Clinical Pharmacology, Medical Faculty, University of Technology, Dresden, Germany